CLINICAL TRIAL: NCT04023656
Title: Prognosis of Paroxysmal Kinesigenic Choreoathetosis in Korea: a Prospective, Observational Study
Brief Title: Prognosis of Paroxysmal Kinesigenic Choreoathetosis in Korea
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han-Joon Kim, Associate Professor, Seoul National University Hospital
Other Study IDs: 1611HJKim808
Record Dates: First submitted 2019-07-12; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Paroxysmal Kinesigenic Choreoathetosis
Keywords: paroxysmal kinesigenic choreoathetosis; Prognosis; Korean population
MeSH Terms: conditions — Familial paroxysmal dystonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the prognosis of paroxysmal kinesigenic choreoathetosis (PKC) in Korean.

DETAILED DESCRIPTION:
PKC is a hyperkinetic movement disorder including dystonia, chorea, athetosis, or ballism, which are characteristically triggered by a sudden movement from rest. The prevalence of this disorder is estimated to be 1 in 150,000 population. Males are more commonly affected than females, and the age of onset is typically in childhood or adolescence. PKC is mainly a familial disorder with autosomal dominant inheritance and incomplete penetrance, but it can occur sporadically. The PRRT2 (proline-rich transmembrane protein 2) gene is believed to be the major causative gene.

The prognosis of PKC is usually favorable. The severity and frequency of the attacks are reduced by anticonvulsant medication such as carbamazepine, and the number of the attacks decreases at the age of 20-30 years. However, there has been little study of long-term prognosis of PKC, and no study has been conducted in Korean population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female PKC patients who were18 years of age and older
* Subjects were diagnosed as paroxysmal kinesigenic choreoathetosis (PKC)
* Subjects were enrolled voluntarily and understood the contents of this trial

Exclusion Criteria:

* Existence of lesions on the brain
* Existence of neurological deficit that suspected lesions on the brain
* Existence of epileptiform discharges on electroencephalogram
* Subjects with secondary PKC which was caused by other disorder or illness
* Existence of illness or problems which made difficult to be enrolled to this trial judged by clinicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators enrolled subjects at the Seoul National University Hospital. Subjects were diagnosed with paroxysmal kinesigenic choreoathetosis (PKC) and followed-up at the Seoul National University Hospital. All subjects were enrolled voluntarily and understood the contents of this trial.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in clinical characteristics of PKC relative to the baseline. | up to 10 years
  Improvement or worsening of the attacks relative to the baseline state assessed by a questionnaire, categorized as following; 1, full remission (absence of the attacks); 2, improvement (more than 50% decreased mean frequency of the attacks); 3, worsening (increased frequency of the attacks).
Changes in clinical characteristics of PKC over the last year. | up to 10 years
  Improvement or worsening of the attacks over the last year assessed by a questionnaire, categorized as following; 1, full remission (absence of the attacks); 2, improvement (more than 50% decreased mean frequency of the attacks); 3, worsening (increased frequency of the attacks).
Changes in medication history of PKC over the last year. | up to 10 years
  Continuation or discontinuation of the medication for relief of the attacks assessed by a questionnaire, categorized as following; 1, continuation of medication; 2, discontinuation of medication.

CONTACTS AND LOCATIONS:
Overall Officials: Han-joon Kim, MD, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mao CY, Shi CH, Song B, Wu J, Ji Y, Qin J, Li YS, Wang JJ, Shang DD, Sun SL, Xu YM. Genotype-phenotype correlation in a cohort of paroxysmal kinesigenic dyskinesia cases. J Neurol Sci. 2014 May 15;340(1-2):91-3. doi: 10.1016/j.jns.2014.02.034. Epub 2014 Mar 3. PMID 24661410
- [Background] Li HF, Chen WJ, Ni W, Wang KY, Liu GL, Wang N, Xiong ZQ, Xu J, Wu ZY. PRRT2 mutation correlated with phenotype of paroxysmal kinesigenic dyskinesia and drug response. Neurology. 2013 Apr 16;80(16):1534-5. doi: 10.1212/WNL.0b013e31828cf7e1. Epub 2013 Mar 27. No abstract available. PMID 23535490
- [Background] Castiglioni C, Lopez I, Riant F, Bertini E, Terracciano A. PRRT2 mutation causes paroxysmal kinesigenic dyskinesia and hemiplegic migraine in monozygotic twins. Eur J Paediatr Neurol. 2013 May;17(3):254-8. doi: 10.1016/j.ejpn.2012.10.010. Epub 2012 Nov 19. PMID 23182655
- [Background] Ebrahimi-Fakhari D, Saffari A, Westenberger A, Klein C. The evolving spectrum of PRRT2-associated paroxysmal diseases. Brain. 2015 Dec;138(Pt 12):3476-95. doi: 10.1093/brain/awv317. Epub 2015 Nov 23. PMID 26598493
- [Background] Bruno MK, Hallett M, Gwinn-Hardy K, Sorensen B, Considine E, Tucker S, Lynch DR, Mathews KD, Swoboda KJ, Harris J, Soong BW, Ashizawa T, Jankovic J, Renner D, Fu YH, Ptacek LJ. Clinical evaluation of idiopathic paroxysmal kinesigenic dyskinesia: new diagnostic criteria. Neurology. 2004 Dec 28;63(12):2280-7. doi: 10.1212/01.wnl.0000147298.05983.50. PMID 15623687
- [Background] Unterberger I, Trinka E. Diagnosis and treatment of paroxysmal dyskinesias revisited. Ther Adv Neurol Disord. 2008 Sep;1(2):4-11. doi: 10.1177/1756285608095119. PMID 21180566
- [Background] Bennett LB, Roach ES, Bowcock AM. A locus for paroxysmal kinesigenic dyskinesia maps to human chromosome 16. Neurology. 2000 Jan 11;54(1):125-30. doi: 10.1212/wnl.54.1.125. PMID 10636137
- [Background] Gardiner AR, Jaffer F, Dale RC, Labrum R, Erro R, Meyer E, Xiromerisiou G, Stamelou M, Walker M, Kullmann D, Warner T, Jarman P, Hanna M, Kurian MA, Bhatia KP, Houlden H. The clinical and genetic heterogeneity of paroxysmal dyskinesias. Brain. 2015 Dec;138(Pt 12):3567-80. doi: 10.1093/brain/awv310. Epub 2015 Nov 23. PMID 26598494
- [Background] Swoboda KJ, Soong B, McKenna C, Brunt ER, Litt M, Bale JF Jr, Ashizawa T, Bennett LB, Bowcock AM, Roach ES, Gerson D, Matsuura T, Heydemann PT, Nespeca MP, Jankovic J, Leppert M, Ptacek LJ. Paroxysmal kinesigenic dyskinesia and infantile convulsions: clinical and linkage studies. Neurology. 2000 Jul 25;55(2):224-30. doi: 10.1212/wnl.55.2.224. PMID 10908896
- [Background] Meneret A, Grabli D, Depienne C, Gaudebout C, Picard F, Durr A, Lagroua I, Bouteiller D, Mignot C, Doummar D, Anheim M, Tranchant C, Burbaud P, Jedynak CP, Gras D, Steschenko D, Devos D, Billette de Villemeur T, Vidailhet M, Brice A, Roze E. PRRT2 mutations: a major cause of paroxysmal kinesigenic dyskinesia in the European population. Neurology. 2012 Jul 10;79(2):170-4. doi: 10.1212/WNL.0b013e31825f06c3. Epub 2012 Jun 27. PMID 22744660
- [Background] Marini C, Conti V, Mei D, Battaglia D, Lettori D, Losito E, Bruccini G, Tortorella G, Guerrini R. PRRT2 mutations in familial infantile seizures, paroxysmal dyskinesia, and hemiplegic migraine. Neurology. 2012 Nov 20;79(21):2109-14. doi: 10.1212/WNL.0b013e3182752ca2. Epub 2012 Oct 17. PMID 23077026